CLINICAL TRIAL: NCT06963125
Title: The Effects of Different Doses of Prune Juice on Bowel Movement Patterns, Constipation Symptoms, and Quality of Life Among Older Adults in Long-Term Care Facilities
Brief Title: The Effects of Prune Juice on Bowel Movement Patterns, Constipation Symptoms, and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: B11304037
Record Dates: First submitted 2025-03-18; First posted 2025-05-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Constipation in Older Adults; Functional Constipation in Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): 30 elderly individuals residing in long-term care facilities, aged between 65 and 100 years, who have been diagnosed with functional constipation.
  Interventions: Dietary Supplement: Low-Dose Prune Juice
- Experimental Group 2 (Experimental): 30 elderly individuals residing in long-term care facilities, aged between 65 and 100 years, who have been diagnosed with functional constipation.
  Interventions: Dietary Supplement: Medium-Dose Prune Juice
- Experimental Group 3 (Experimental): 30 elderly individuals residing in long-term care facilities, aged between 65 and 100 years, who have been diagnosed with functional constipation.
  Interventions: Dietary Supplement: High-Dose Prune Juice

INTERVENTIONS:
Dietary Supplement: Low-Dose Prune Juice — Intervention Name: Prune Juice 100 mL/day Description: 100 mL prune juice daily (1.07 g dietary fiber), administered once each morning for 4 weeks.
  Arms: Experimental Group 1
Dietary Supplement: Medium-Dose Prune Juice — Intervention Name: Prune Juice 150 mL/day Description: 150 mL prune juice daily (1.61 g dietary fiber), administered once each morning for 4 weeks.
  Arms: Experimental Group 2
Dietary Supplement: High-Dose Prune Juice — Intervention Name: Prune Juice 200 mL/day Description: 200 mL prune juice daily (3.22 g dietary fiber), administered once each morning for 4 weeks.
  Arms: Experimental Group 3

SUMMARY:
This study investigates the effects of different prune juice dosages on bowel movement patterns, constipation symptoms, and quality of life in older adults. Using a factorial experimental design, 90 participants aged 65 to 100 with functional constipation will be randomly assigned to receive 100 mL, 150 mL, or 200 mL of prune juice daily for four weeks. The study aims to determine a safe and effective dosage for constipation management, offering a non-pharmacological approach to improving bowel health in older adults.

DETAILED DESCRIPTION:
Constipation is a prevalent issue among older adults, leading to physical discomfort and long-term health complications. Non-pharmacological interventions are essential for effective management. This study aims to compare the effects of different prune juice dosages on bowel movement patterns, constipation symptoms, and quality of life to determine a safe and effective dosage for older adults. A factorial experimental design will be employed, with 90 participants aged 65 to 100 who are conscious, able to express their opinions, and diagnosed with functional constipation. Participants will be randomly assigned to three groups receiving 100 mL, 150 mL, or 200 mL of prune juice daily for four weeks. The outcomes will be assessed at five time points: before the intervention (T0), after one week (T1), after two weeks (T2), after three weeks (T3), and after four weeks (T4).

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65 to 100 years
* Cognitively aware and able to express their opinions
* Diagnosed with functional constipation

Exclusion Criteria:

* Diagnosis of diabetes mellitus
* Cognitive impairment, including moderate to severe dementia or psychiatric disorders
* Aphasia
* Severe hearing impairment
* Presence of gastrointestinal diseases, including:
* Gastrointestinal bleeding
* Intestinal obstruction
* Abdominal tumors
* Irritable bowel syndrome
* Acute diverticulitis
* Diarrhea
* Crohn's disease
* Ulcerative colitis
* History of abdominal surgery
* Regular use of probiotics
* Regular use of traditional Chinese medicine or folk remedies for constipation relief
* Difficulty swallowing or risk of aspiration
* Major illnesses, such as current cancer treatment or severe cardiovascular diseases
* Currently hospitalized

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Stool Consistency Measured by Bristol Stool Form Scale (BSFS) | From study enrollment to the end of the 4-week intervention
  Stool consistency will be assessed using the Bristol Stool Form Scale (BSFS), a 7-point scale that classifies stool into 7 types: Type 1 = separate hard lumps Type 7 = entirely liquid Types 3 to 5 are considered normal. The mean change in BSFS score from baseline to Week 4 will be measured. Higher or lower scores reflect changes in stool consistency severity.
Change in Constipation Symptoms Measured by PAC-SYM | From study enrollment to the end of the 4-week intervention
  Constipation symptoms will be assessed using the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire. This instrument includes 12 items across abdominal, stool, and rectal symptom subscales. Each item is rated from 0 (no symptoms) to 4 (very severe). The total score ranges from 0 to 48, with higher scores indicating worse symptoms. The change in total PAC-SYM score from baseline to Week 4 will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Licensed Long-Term Care Institutions in Chiayi Region, Chiayi City, Chiayi County, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the absence of a data-sharing infrastructure at this time.